CLINICAL TRIAL: NCT02467426
Title: Isolated Thoracic Perfusion With Hemofiltration (ITP-F) for Pretreated and Progressive Malignant Pleural Mesothelioma
Brief Title: Isolated Thoracic Perfusion (ITP-F) for MPM
Status: Completed | Type: Observational
Sponsor: Medias Klinikum for Surgical Oncology (Other)
Responsible Party: Principal Investigator, Prof. Andreas Sendler, Senior Consultant, Dept. of Surgical Oncology, Medias Klinikum for Surgical Oncology
Other Study IDs: 0001
Record Dates: First submitted 2015-05-26; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Mesothelioma
Keywords: Mesothelioma, malignant; Chemotherapy
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Drug Therapy; Mitoxantrone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemotherapy: intraarterial chemotherapy with cisplatin and mitoxantrone
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — intraarterial infusion of cisplatin and mithoxantrone
  Other Names: CDDP; Mitoxantrone

SUMMARY:
This is an observational study of isolated thoracic perfusion with subsequent hemofiltration to lower the concentration of the cytotoxic drugs as a locoregional therapeutic strategy in malignant pleural mesothelioma.

DETAILED DESCRIPTION:
Treatment of patients with progressive malignant pleural mesothelioma (MPM) after multimodal therapy is a therapeutic challenge. Survival of the patients is low and the treatment options are sparse. This is an observational study of isolated thoracic perfusion with subsequent hemofiltration as a locoregional therapeutic strategy in this situation.

23 pts. with epithelioid MPM were included in this phase II study after informed consent. All patients had progressive disease after multiple therapies and were recommended BSC of a MDT. Following insertion of a venous and arterial 21 ch. stop flow catheter via a femoral access, the inferior vena cava was blocked beneath the right atrium, the arterial catheter was blocked in the aorta at the diaphragm. The upper arms were blocked by pneumatic cuffs. Chemotherapy was given via the arterial catheter. Chemotherapy consisted of 60mg/m2 cisplatinum and 15mg/m2 mitoxantrone q for 3 weeks until progress. After administration of chemotherapy, thoracic perfusion with blocked stop-flow catheters was maintained for 15 minutes. After de-blocking of the catheters, hemofiltration was performed for 45 min. with 5l filtrate. The endpoint of the study was overall survival.Secondary endpoint was toxicity.

ELIGIBILITY:
Inclusion Criteria:

* History of pre-treated Malignant Pleural Mesothelioma, Progress after Staging

Exclusion Criteria:

* Drug abuse, distant metastases, no bone marrow function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with progressive malignant mesothelioma after failure of convetional multimodal therapy including resection
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Survival | one year survival
  Kaplan-Maier Plot

SECONDARY OUTCOMES:
Toxicity | 4 weeks after therapy
  Toxicity was measured by Common Toxicity Criteria Vers. 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Karl R. Aigner, MD, Principal Investigator — Medias Klinikum Burghausen

REFERENCES:
- See also: homepage of the hospital — http://www.medias-klinikum.de